CLINICAL TRIAL: NCT03708757
Title: Comparison Of PIR Technique With Eccentric Isotonic Muscle Contraction on Hamstring Spasticity in CP Child
Brief Title: Effect of Post Isometric Relaxation Technique & Eccentric Muscle Contraction on Hamstring Spasticity in CP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Shafaq Bano
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Spastic Cerebral Palsy
Keywords: Cerebral palsy; Post Isometric Relaxation; Hamstring Spasticity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Experimental Study
Who Masked: Participant
Masking Description: This will be a single blinded study.Participants will be randomly allocated to PIRT Group (I) or EMET Group (II)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post isometric relaxation - Group I (Experimental): Group I will receive post isometric relaxation techniques in order to reduce hamstring spasticity. This technique induces relaxation and decreases spasticity in muscles
  Post isometric relaxation (3 sets of 10 repetitions ,1 session in a day, 30 minutes, 4 days a week for 6 weeks.) Stretching Exercises (10 reps 3sets) hold for 2 sec
  Interventions: Other: Post isometric relaxation - Group I
- Eccentric Muscle contraction - Group II (Active Comparator): Eccentric Muscle contraction lengthens the spastic muscles and enhance joint flexibility.
  Hot Pack for (10 MINTS) Eccentric stretching (3 sets of 10 repetitions ,1 session in a day, 30 minutes, 4 days a week for 6 weeks.) Stretching Exercise(10 reps 3sets) hold for 2 sec In both experimental groups PIR and Eccentric stretching is applied on hamstring to
  Interventions: Other: Eccentric Muscle contraction - Group II

INTERVENTIONS:
Other: Post isometric relaxation - Group I — Post isometric relaxation (PIR) techniques are used by orthopedic manual physical therapists to enhance the flexibility of muscles and to increase the joint range of motion
  Arms: Post isometric relaxation - Group I
Other: Eccentric Muscle contraction - Group II — and Eccentric muscle energy techniques(EME) techniques are used by orthopedic manual physical therapists to enhance the flexibility of muscles and to increase the joint range of motion
  Arms: Eccentric Muscle contraction - Group II

SUMMARY:
Cerebral Palsy is a disorder of movement and posture due to deficit or lesion of immature brain. Out of all types of cerebral palsy 77.4% is spastic cerebral palsy. Spasticity is resistance to externally imposed movement increases with increasing speed of stretch and varies with the direction of joint movement. In this research the aim of our study is to measure the effects of post isometric relaxation and eccentric muscle energy technique of spasticity of hamstring muscle in cerebral palsy children in randomized controlled study. Study duration is of six months. Sampling will be lottery method. Inclusion criteria will include individuals having age between five to fifteen with diplegic cerebal palsy, well oriented and spastic hamstrings with Ashworth score +2 or +3.Exclusion criteria includes children with flaccid and mixed cerebral palsy, quadriplegic and hemiplegic cerebral palsy and mentally retarded. Data will be collected on structured questionnaire. those individuals who fulfill inclusion criteria will be divided into two groups .both groups will be treated with hot packs for ten minutes and static stretching. Group 1 will be given post isometric relaxation technique and group 2 will be given eccentric muscle energy technique. Post interventional analysis will be done at sixth week. Data will be analysed with SPSS 21.

DETAILED DESCRIPTION:
The primary purpose of this study is to investigate effects of eccentric isotonic contraction on on hamstring flexibility of cerebral palsy children,and to investigate effects of post isometric relaxation on on hamstring flexibility of cerebral palsy children.It is a randomized control trial. this study will be conducted in PAF School for PSN Norkhan base Rawalpindi. Data collection time is from Oct 2018- March 2019. Sample size is 30 CP child,15 in each group calculated by Open Epi Tool.

Ap per Inclusion criteria only those participants will be included with age bracket 5-15 years,spastic diplegic , well oriented and on modified Ashworth scale their score is +2 or +3. Children with flaccid and mixed cerebral palsy,Quadriplegic and hemiplegic cerebral palsy or Mentally retarded will not be part of study. Those patients who fulfill inclusion criteria are divided in to two groups. Intervention will be provided and Assessments should be done on 1st on baseline and then after 6 weeks.Data Collection Tools will be Gross Motor Functional scale,Goniometry for measuring joint ranges and Motor Assessment Scale for measuring their functional status.

ELIGIBILITY:
Inclusion Criteria:

* Children with spastic cerebral palsy
* Diplegic cerebral palsy
* well oriented
* Spastic hamstrings with Ashworth score +2 or +3

Exclusion Criteria:

* Children with flaccid and mixed cerebral palsy
* Quadriplegic and hemiplegic cerebral palsy
* Mentally retarded

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Goniometry | 6th week
  change from baseline.This tool is used to measure range of motion of hip joint and knee joint

SECONDARY OUTCOMES:
Gross motor Functional Scale | 6th week
  Change from baseline.Tool is used to measure the functional status of patients. The Gross Motor Function Classification System (GMFCS) for cerebral palsy is based on self-initiated movement, with emphasis on sitting, transfers, and mobility. It gives information about levels of limitations.
  LEVEL I - Walks without Limitations LEVEL II - Walks with Limitations LEVEL III - Walks Using a Hand-Held Mobility Device LEVEL IV - Self-Mobility with Limitations; May Use Powered Mobility LEVEL V - Transported in a Manual Wheelchair

CONTACTS AND LOCATIONS:
Overall Officials: imran Amjad, Principal Investigator — Associate Professor
Locations (2):
- Pakistan (2):
  - Imran Amjad, Islamabad, Punjab Province
  - Riphah International University, Islamabad

REFERENCES:
- [Background] Czaprowski D, Leszczewska J, Kolwicz A, Pawlowska P, Kedra A, Janusz P, Kotwicki T. The comparison of the effects of three physiotherapy techniques on hamstring flexibility in children: a prospective, randomized, single-blind study. PLoS One. 2013 Aug 12;8(8):e72026. doi: 10.1371/journal.pone.0072026. eCollection 2013. PMID 23951281
- [Background] Smith M, Fryer G. A comparison of two muscle energy techniques for increasing flexibility of the hamstring muscle group. J Bodyw Mov Ther. 2008 Oct;12(4):312-7. doi: 10.1016/j.jbmt.2008.06.011. Epub 2008 Aug 6. PMID 19083689
- [Background] Lee GP, Ng GY. Effects of stretching and heat treatment on hamstring extensibility in children with severe mental retardation and hypertonia. Clin Rehabil. 2008 Sep;22(9):771-9. doi: 10.1177/0269215508090067. PMID 18728130
- [Background] Adel Rashad ahmed , A comparative study of muscle energy technique and dynamic stretching on hamstring flexibility. Bulletin of faculty of physical therapy.2011;16(1)
- [Background] Reid S, Hamer P, Alderson J, Lloyd D. Neuromuscular adaptations to eccentric strength training in children and adolescents with cerebral palsy. Dev Med Child Neurol. 2010 Apr;52(4):358-63. doi: 10.1111/j.1469-8749.2009.03409.x. Epub 2009 Sep 8. PMID 19737297